CLINICAL TRIAL: NCT00750828
Title: Gingival Wetness and Gingival Crevicular Fluid Volume in Patients With Dry Mouth
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Burak Demiralp, Hacettepe University Faculty of Dentistry Department of Periodontology
Other Study IDs: Hacettepe # FON 03/6-14
Record Dates: First submitted 2008-09-10; First posted 2008-09-11 (Estimated); Last update posted 2008-09-11 (Estimated); Status verified 2008-09

CONDITIONS: Xerostomia; Sjogren's Syndrome
Keywords: Saliva; Sjögren's Syndrome; GCF; Oral Mucosal Wetness
MeSH Terms: conditions — Xerostomia; Sjogren's Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The investigators questioned whether patients with dry mouth complaints display any reduction in residual saliva coating the gingiva and other selected mucosal surfaces. We further intended to test the hypothesis that Gingival Crevicular Fluid volume in patients with dry mouth could be different from that of control subjects. Correlations between gingival/mucosal wetness; and unstimulated whole salivary flow rate or minor salivary gland secretion rates and the correlations between clinical periodontal status and salivary measures were also attempted.

ELIGIBILITY:
Inclusion Criteria:

* For test group dry mouth complaints and with a diagnosis ofSjogren's Syndrome

Exclusion Criteria:

* Other medical problems that effect salivary glands

Ages: 46 Years to 56 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: The data for this study were taken from 28 subjects at the Department of Periodontology, Hacettepe University from 2004 to 2007. The study group consisted of 14 patients with dry mouth complaints. All of them had the diagnosis of Sjögren's syndrome and ten of them were on therapy for sicca symptoms.
  Fourteen randomly selected age-matched systemically healthy females were also included as a control group
Sampling Method: Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2004-01; Primary Completion 2007-12 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Burak Demiralp, DDS PhD, Study Director — Hacettepe University Faculty of Dentistry Department of Periodontology
Locations (1):
- Department of Periodontology, Faculty of Dentistry, Hacettepe University,, Ankara, Turkey (Türkiye)